CLINICAL TRIAL: NCT05037643
Title: Pre-emptive Transjugular Intrahepatic Portosystemic Shunt (TIPS) in Pediatric Patients With Cystic Fibrosis Related Liver Disease and Non-cirrhotic Portal Hypertension
Brief Title: Pre-emptive Transjugular Intrahepatic Portosystemic Shunt (TIPS) in Cystic Fibrosis Related Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B67020071504
Record Dates: First submitted 2021-08-16; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis Liver Disease; Portal Hypertension Due to Cystic Fibrosis (Disorder); Portal Hypertension, Noncirrhotic
Keywords: Transjugular Intrahepatic Portosystemic Shunt; Gastrointestinal bleeding; Hypersplenism
MeSH Terms: conditions — Hypertension, Portal; Gastrointestinal Hemorrhage; Hypersplenism | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Intervention Model Description: Prospective single-arm study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-emptive TIPS in Cystic Fibrosis Related Liver Disease and non-cirrhotic portal hypertension (Experimental): Patients with CFLD without cirrhosis were eligible for a pre-emptive TIPS, when early (asymptomatic) signs of portal hypertension. All procedures were performed under general anaesthesia by an experienced interventional radiologist. Depending on the patient's age and physiognomy, TIPS was created following a conventional transjugular technique as for adults or by a dedicated combined percutaneous transhepatic-transjugular (PIPS) approach for small children. Routinely, an expanded polytetrafluoroethylene-covered endoprosthesis was used for shunt creation. If the sheath could not be negotiated into the main portal vein, a self-expandable, non-covered stent was placed. We did not pursue a minimum gradient reduction.
  Percutaneous liver biopsy was performed during TIPS procedure to confirm the diagnosis of fibrosis or cirrhosis.
  Interventions: Procedure: TIPS

INTERVENTIONS:
Procedure: TIPS — Transjugular Intrahepatic Portosystemic Shunt is performed to prevent / treat symptomatic portal hypertension

SUMMARY:
Portal hypertension (PHT) and its sequelae are the most clinically important manifestation in cystic fibrosis related liver disease (CFLD), with end-stage liver failure as a late and rare manifestation. The aim is to evaluate the safety and efficacy of a pre-emptive Transjugular Intrahepatic Portosystemic Shunt (TIPS) for the prophylaxis of variceal bleeding in pediatric CFLD patients with subclinical non-cirrhotic portal hypertension (NCPH)

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most frequent autosomal recessive disorder in Caucasians caused by a mutation in the cystic fibrosis transmembrane conductance regulator gene. Cystic Fibrosis associated Liver Disease (CFLD) is a well-known complication and includes a wide range of hepatobiliary diseases. The clinical outcome in CFLD is largely determined by PHT and its sequelae. Variceal bleeding is the most feared complication. Currently, there is no medical therapy to delay or reverse clinically established CFLD.Treatment focuses on screening for and managing the complications of portal hypertension and optimizing nutritional status. Eventually, liver transplantation (LT) is an effective therapeutic option for CF patients with end-stage liver failure, treatment resistant, and complicated portal hypertension.

TIPS placement is a well-established procedure for portal vein decompression in adults. In retrospective case studies of severe CFLD cirrhosis in pediatric populations, TIPS has been proven a feasible option in acute or refractory variceal bleeding and as a bridge to LT. In CFLD patients, little data are available on the long-term outcome of treatments to mitigate PHT. In this trial, the primary aim was to evaluate the safety and efficacy of a pre-emptive TIPS for the prophylaxis of variceal bleeding in non-cirrhotic CFLD with early PHT. The secondary aim was to investigate the long-term clinical outcome of a pre-emptive TIPS and in more particular, whether TIPS might effectively postpone LT.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis
* Liver disease detected by an abnormal physical examination (hepatomegaly or splenomegaly, confirmed on US), abnormalities of liver function tests (increase of AST, ALT, GGT levels above the upper normal limits) or ultrasonographic evidence of liver involvement (US liver score ≥ 5).
* Indirect signs of portal hypertension on Doppler US
* Progressive portal hypertension / liver disease on bi-monthly follow-up, evaluated by physical examination, blood analysis and US

Exclusion Criteria:

* Cirrhosis on biopsy
* Symptomatic portal hypertension (Portosytemic pressure gradient > 10 mmHg)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Variceal bleeding | Through study completion, an average of 10 year
  Variceal bleeding, diagnosed on endoscopy, is regarded as the main complication of portal hypertension from cystic fibrosis liver disease

SECONDARY OUTCOMES:
Hypersplenism | Through study completion, an average of 10 year
  Thrombocytopenia causes an increased bleeding tendency. Increasing splenomegaly causes earlier concerns with abdominal distension and decreased appetite by gastric compression. In symptomatic hypersplenism, a surgical splenorenal shunt or splenectomy might be indicated.

OTHER OUTCOMES:
Liver transplant/splenectomy-free survival | Through study completion, an average of 10 year
  Transplant/splenectomy-free survival time was calculated from date of TIPS to the following event: transplant, splenectomy and death from any cause.
Model for end-stage liver disease (MELD) score | Through study completion, an average of 10 year
  The Model for End-Stage Liver Disease, or MELD, is a scoring system for assessing the severity of chronic liver disease.
Body Mass Index (BMI) for age Z-score | Through study completion, an average of 10 year
  BMI-for age Z-scores are measures of relative weight adjusted for child age and sex defined by the Flemish growth charts
Length for age Z-score | Through study completion, an average of 10 year
  Length-for age Z-scores are measures of relative length adjusted for child age and sex defined by the Flemish growth charts

CONTACTS AND LOCATIONS:
Overall Officials: Luc Defreyne, M.D., Ph.D, Principal Investigator — University Ghent Hospital

IPD SHARING:
Plan to Share IPD: No